CLINICAL TRIAL: NCT05677165
Title: The Relationship Between Driving Pressure, Mechanical Power, Oxygenation and Saturation Indices: Retrospective Observational Study
Status: Completed | Type: Observational
Sponsor: Bakirkoy Dr. Sadi Konuk Research and Training Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021/293
Record Dates: First submitted 2022-11-21; First posted 2023-01-10 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2022-12

CONDITIONS: Acute Respiratory Distress Syndrome; Pneumonia
Keywords: acute respiratory distress syndrome; pneumonia; oxygenation index; saturation index
MeSH Terms: conditions — Respiratory Distress Syndrome; Pneumonia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
By using Mechanical Power and Driving Pressure instead of Pmean we calculate new oxygen saturation indices like Driving Pressure Oxygen Index (OIDP), Dynamic Power Oxygen Index (OIMPdyn), Total Power Oxygen Index (OIMPtot), Driving Pressure Saturation Index (OSIDP), Dynamic Power Saturation Index (OSIMPdyn) ve Power Saturation Index (OSIMPtot).

New oxygenation and saturation indices are able to predict ICU mortality better than the conventional indexes and rates.

ELIGIBILITY:
Inclusion Criteria:

- Patients with a diagnosis of Covid-19 related Acute Respiratory Syndrome (C-ARDS) which hospitalized in Bakirköy Dr. Sadi Konuk Training and Research Hospital intensive care unit

Exclusion Criteria:

* Patients who did not receive invasive mechanical ventilation support.
* Patients who stayed in the intensive care unit for less than 24 hours.
* Patients with missing data
* Patients who received mechanical ventilation support for less than 24 hours
* Patients with Chronic Obstructive Pulmonary Disease (COPD).
* Patients with congestive heart failure
* Patients who underwent tube thoracostomy due to tension pneumothorax
* Patients who received Extracorporeal Membrane Oxygenation (ECMO) support

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The data of 784 patients with a diagnosis of Covid-19 hospitalized in the 28-bed intensive care unit of the Bakirkoy Dr. Sadi Konuk Training and Research Hospital were obtained by using structured query language (sql) queries from the 'ImdSoft-Metavision/QlinICU Clinical Decision Support (Israel) system'.173 patients who did not receive invasive mechanical ventilation support, 64 patients who stayed in the intensive care unit for less than 24 hours, 40 patients with missing data, and 38 patients who received mechanical ventilation support for less than 24 hours were excluded from the study.24 patients with COPD, 27 patients with congestive heart failure, and 11 patients who underwent tube thoracostomy due to tension pneumothorax were excluded from the study.In addition, 46 patients who received ECMO support were excluded from the study due to the possibility that ECMO may have an effect on respiratory variables. The remaining 361 patients were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 361 (Actual)
Dates: Start 2020-03-18 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-28 (Actual)

PRIMARY OUTCOMES:
In hospital mortality | 28 days
  we estimate hospital mortality mortality by calculating new oxygenation index

SECONDARY OUTCOMES:
Mechanical ventilatory free days | 30 days
  we estimate hospital mortality mortality by calculating new saturation index

CONTACTS AND LOCATIONS:
Locations (1):
- Bakirköy Dr sadi konuk Education hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided